CLINICAL TRIAL: NCT00627250
Title: Utility of Amantadine Hydrochloride in the Treatment of Post-traumatic Irritability: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Utility of Amantadine Hydrochloride in the Treatment of Post-traumatic Irritability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-02-06A; H133A020522
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2008-02

CONDITIONS: Irritable Mood; Aggression; Traumatic Brain Injury
Keywords: Irritability; Aggression; Brain Injury; Amantadine; Irritability and Aggression Due to Traumatic Brain Injury
MeSH Terms: conditions — Aggression; Brain Injuries, Traumatic; Brain Injuries | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Amantadine 100 mg every morning and 12 noon
  Interventions: Drug: Amantadine
- B (Placebo Comparator): Placebo tablet every morning and 12 noon
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — Amantadine 100 mg every morning and 12 noon
  Other Names: Symmetrel

SUMMARY:
The purpose of this study is to determine if amantadine hydrochloride given 100 mg in the morning and at noon is safe and effective in the treatment of mood and behavior changes (i.e. irritability) after sustaining traumatic brain injury.

DETAILED DESCRIPTION:
Amantadine hydrochloride is a drug used commonly in clinical practice at the Carolinas Rehabilitation for the treatment of mood and behavior changes following traumatic brain injury. Clinical observation suggests that the use of amantadine improves caregiver report of "irritability" though there are no studies to validate this observation. This study investigates the efficacy and side effect profile of amantadine hydrochloride given in 2 doses of 100 mgs each. Subjects are screened during regularly scheduled clinic appointments for the presence of irritability. If they are interested in possible participation in the study, they will be invited to meet with the research coordinator who will obtain informed consent. If the subject meets all the inclusion/exclusion requirements, they will leave clinic with study medication and begin taking the drug the next day. There will be a safety call between day 3 and 5 where the dose may be reduced to once per day. Follow-up assessment occurs at day 14 (by phone) and day 28 (in clinic). At study completion, the subject will have the opportunity to receive a prescription for amantadine as part of ongoing clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Closed head injury (defined as brain injury or impaired brain function resulting from externally inflicted trauma without penetrating injury) at least 6 months prior to enrollment.
* Age at time of enrollment: 16 - 65 inclusive (i.e., on or after 16th birthday, up to day before 66th birthday).
* Voluntary informed consent of patient and informant.
* Subject and informant willing to comply with the protocol, & are available for all scheduled clinic visits.
* Neuropsychiatric Inventory (NPI) Irritability Domain score > 2.
* Medically and neurologically stable during the month prior to enrollment.
* If taking antidepressant, anxiolytic, hypnotic, or stimulant medications, no change anticipated in these medications during the month prior to enrollment.
* No change in therapies or medications planned during the 28-day participation.
* No surgeries planned during the 28-day participation.
* Vision, hearing, speech, motor function, and comprehension must be sufficient for compliance with all testing procedures. Ability to interact and verbalize sufficient to participate in assessments.
* Informant (family member or close friend) who lives with the participant with daily interaction in order to observe occurrences of irritability.

Exclusion Criteria:

* Patients without a reliable informant
* Penetrating head injury
* Injury < 6 months prior to enrollment
* Inability to interact sufficient for communication with caregiver
* Acute and rehabilitation records unavailable or incomplete
* DSM-IV diagnosis of schizophrenia or psychosis
* Diagnosis of progressive or additional neurologic disease (such as, Alzheimer's disease, parkinson's disease, multi-infarct dementia, other cerebrovascular disorders with dementia, prior cerebrovascular accident, Huntington's disease, olivopontocerebellar atrophy, multisystem atrophy, multiple sclerosis, ALS, CNS tumor, progressive supranuclear palsy).
* Diagnosis of seizure in the month prior to enrollment.
* Previous allergy or adverse reaction to study drug
* Ingestion of amantadine hydrochloride during the month prior to enrollment.
* Concomitant use of neuroleptic agents or phenelzine
* Creatinine clearance <60
* Pregnancy (Beta-HCG performed on all females of child-bearing potential) and lactating females.
* Clinical signs of active infection

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2003-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (Irritability Domain frequency and severity) | 28 days

SECONDARY OUTCOMES:
Neuropsychiatric Inventory Irritability and Aggression(Caregiver distress scores) | 28 days
Neuropsychiatric Inventory Aggression Domain (frequency and severity) | 28 days
Global Impression of Change rated by clinician, individual with brain injury and caregiver | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Flora M Hammond, M.D., Principal Investigator — Carolinas Rehabilitation

REFERENCES:
- [Background] Gualtieri T, Chandler M, Coons TB, Brown LT. Amantadine: a new clinical profile for traumatic brain injury. Clin Neuropharmacol. 1989 Aug;12(4):258-70. No abstract available. PMID 2680078
- [Background] HERRMANN EC Jr, GABLIKS J, ENGLE C, PERLMAN PL. Agar diffusion method for detection and bioassay of antiviral antibiotics. Proc Soc Exp Biol Med. 1960 Mar;103:625-8. doi: 10.3181/00379727-103-25617. No abstract available. PMID 14401357
- [Background] Schwab RS, England AC Jr, Poskanzer DC, Young RR. Amantadine in the treatment of Parkinson's disease. JAMA. 1969 May 19;208(7):1168-70. No abstract available. PMID 5818715
- [Background] Beers SR, Skold A, Dixon CE, Adelson PD. Neurobehavioral effects of amantadine after pediatric traumatic brain injury: a preliminary report. J Head Trauma Rehabil. 2005 Sep-Oct;20(5):450-63. doi: 10.1097/00001199-200509000-00006. PMID 16170253
- [Background] Gianutsos G, Chute S, Dunn JP. Pharmacological changes in dopaminergic systems induced by long-term administration of amantadine. Eur J Pharmacol. 1985 Apr 16;110(3):357-61. doi: 10.1016/0014-2999(85)90564-3. PMID 2861102
- [Background] Aoki FY, Sitar DS. Clinical pharmacokinetics of amantadine hydrochloride. Clin Pharmacokinet. 1988 Jan;14(1):35-51. doi: 10.2165/00003088-198814010-00003. PMID 3280212
- [Background] Allen RM. Role of amantadine in the management of neuroleptic-induced extrapyramidal syndromes: overview and pharmacology. Clin Neuropharmacol. 1983;6 Suppl 1:S64-73. doi: 10.1097/00002826-198300061-00009. No abstract available. PMID 6196112
- [Background] Stone TW. Evidence for a non-dopaminergic action of amantadine. Neurosci Lett. 1977 May;4(6):343-6. doi: 10.1016/0304-3940(77)90181-1. PMID 19556187
- [Background] Weller M, Kornhuber J. A rationale for NMDA receptor antagonist therapy of the neuroleptic malignant syndrome. Med Hypotheses. 1992 Aug;38(4):329-33. doi: 10.1016/0306-9877(92)90027-a. PMID 1337136
- [Background] Riederer P, Lange KW, Kornhuber J, Danielczyk W. Pharmacotoxic psychosis after memantine in Parkinson's disease. Lancet. 1991 Oct 19;338(8773):1022-3. doi: 10.1016/0140-6736(91)91888-2. No abstract available. PMID 1681331
- [Background] Edby K, Larsson J, Eek M, von Wendt L, Ostergard B. Amantadine treatment of a patient with anoxic brain injury. Childs Nerv Syst. 1995 Oct;11(10):607-9. doi: 10.1007/BF00301001. PMID 8556729
- [Background] Chandler MC, Barnhill JL, Gualtieri CT. Amantadine for the agitated head-injury patient. Brain Inj. 1988 Oct-Dec;2(4):309-11. doi: 10.3109/02699058809150901. PMID 3203176
- [Background] Rosati DL. Early polyneuropharmacologic intervention in brain injury agitation. Am J Phys Med Rehabil. 2002 Feb;81(2):90-3. doi: 10.1097/00002060-200202000-00003. PMID 11807342
- [Background] Shiller AD, Burke DT, Kim HJ, Calvanio R, Dechman KG, Santini C. Treatment with amantadine potentiated motor learning in a patient with traumatic brain injury of 15 years' duration. Brain Inj. 1999 Sep;13(9):715-21. doi: 10.1080/026990599121269. PMID 10507453
- [Background] Schneider WN, Drew-Cates J, Wong TM, Dombovy ML. Cognitive and behavioural efficacy of amantadine in acute traumatic brain injury: an initial double-blind placebo-controlled study. Brain Inj. 1999 Nov;13(11):863-72. doi: 10.1080/026990599121061. PMID 10579658
- [Background] Van Reekum R, Bayley M, Garner S, Burke IM, Fawcett S, Hart A, Thompson W. N of 1 study: amantadine for the amotivational syndrome in a patient with traumatic brain injury. Brain Inj. 1995 Jan;9(1):49-53. doi: 10.3109/02699059509004571. PMID 7874096
- [Background] Zafonte RD, Watanabe T, Mann NR. Amantadine: a potential treatment for the minimally conscious state. Brain Inj. 1998 Jul;12(7):617-21. doi: 10.1080/026990598122386. PMID 9653525
- See also: Related Info — http://www.carolinasrehabilitation.org/